CLINICAL TRIAL: NCT03691233
Title: Clinical Audit on Diagnosis and Management of Neonatal Shock
Brief Title: Diagnosis and Management of Neonatal Shock
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Walaa Ahmed Ezzat Sadak, Principal investigator, Assiut University
Other Study IDs: neonatal shock
Record Dates: First submitted 2018-09-19; First posted 2018-10-01 (Actual); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Neonatal Disorder
MeSH Terms: conditions — Infant, Newborn, Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Clinical audit on diagnosis and management of neonatal shock — intervenous
  Other Names: fliuds

SUMMARY:
The aim of this clinical audit is to assess the degree of adherence of medical physicians in Assiut university children hospital protocol for diagnosis and management of neonatal shock to the international guidelines.

DETAILED DESCRIPTION:
Introduction Shock is defined as a state of impaired cellular energy (ATP) synthesis when tissue oxygen delivery no longer satisfies tissue oxygen demand (Kleinman etal., 2012)

Shock is an independent predictor of early neonatal mortality and more often a problem in preterm infants than in term infants, even late preterm infants are at much higher risk (Femitha and Bhat, 2012)

In the first phase of shock, perfusion and oxygen delivery is maintained towards the so-called vital organs (heart, brain, and adrenal glands) by selective regional vasodilation in combination with vasoconstriction to non-essential tissues, such as muscles, skin, kidneys, and the splanchnic tissues. This is the compensated stage of shock. As the product of cardiac output (which falls) and systemic vascular resistance (which increases), blood pressure actually remains in the normal range in a compensated shock. When this redistribution fails, perfusion and oxygenation of the vital organs will become impaired, resulting in multi-organ dysfunction. In this phase of uncompensated shock, systemic hypotension might be expected (Willem etal., 2018)

Echocardiography is one of the emerging technologies that can be used to measure cardiac output in critically ill newborn infants, especially since the clinical estimation of cardiac output is rather inaccurate (de Boode, 2010)

Diagnosis of Shock

The clinical diagnosis of shock in the early compensated phase often depends on assessment of peripheral perfusion,pulse volume, heart rate changes, metabolic acidosis and urine output.

Ideally, shock should be diagnosed at this stage. In the later uncompensated phase, blood pressure (BP) becomes a key parameter for monitoring and for titrating inotropes and fluids Willem etal.,2018). )

Clinicians rely on BP measurements to diagnose hypotension and to titrate therapy. Hypotension in preterm infants has been associated with an increased risk of intraventricular hemorrhage (Vishnu and Plakkal, 2015)

Treatment of Shock:

1. Volume Expanders

   It is common practice to give one or two normal saline boluses when neonates present in shock, before assessing the need for inotropes.

   Apart from saline, albumin or other colloids are also sometimes used for volume expansion.
2. Drug Therapy of Neonatal Shock

Dopamine is an endogenous catecholamine and has been shown to raise the blood pressure in hypotensive infants better than either albumin or dobutamine (Osborn and Evan, 2005) Cardiac arrhythmias And extravasation injury are potential adverse effects (Osborn etal., 2004)

Dobutamine, unlike dopamine, does not have endocrine effects and does not depend on the release of endogenous catecholamines for effect. It is predominantly inotropic, with some vasodilator effects, Indeed, there is some evidence that dobutamine is better than dopamine at increasing and maintaining systemic blood flow in preterm infants with low systemicblood flow (Subhedar and Shaw, 2003).

Epinephrine is usually used when shock is refractory to dopamine and dobutamine, although some use it as a first line drug, especially when septic shock is suspected (Maria etal., 2004)

Norepinephrine use in neonates is uncommon due to its vasoconstrictive effects, resulting in organ hypoperfusion and increased myocardial work (Pierre etal., 2008)

Hydrocortisone is most commonly used in catecholamine resistant shock in treatment of hypotension in very low birth weight infants (vishnu and plakkal, 2015). Hyperglycemia can be a troublesome short-term side effect (Ng etal., 2006)

Vasopressin is a potent vasoconstrictor and useful in vasodilatory shock (Brierley etal., 2009).

Supportive Treatment:

Pulmonary Support. Most neonates with shock requiring inotropic support will also require mechanical ventilation.(especially <28 wk) (Saugstad and Aune, 2014].

Antibiotics.

* Empirical antibiotics should be chosen based on prevailing infection patterns in each NICU (Adrienne etal., 2003)

Newer Developments in the Management of Neonatal Shock

Milrinone and amrinone are phosphodiesterase III inhibitors. they are vasodilators, hypotension can result. However, they are excellent inotropes and can also reduce pulmonary pressures (Nick etal., 2009)

Levosimendan is a newer drug which causes vasodilatation and improves calcium coupling to troponin, resulting in an increase in myocardial contractility (Papoff etal., 2012)

ELIGIBILITY:
Inclusion Criteria:

* All neonates (preterm or full term) who are developing shock

Exclusion Criteria:

* Neonates with multiple congenital anomalies

Ages: 1 Minute to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The neonates who are admitted to neonatology Unit at Assiut University Children Hospital through this period
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2019-10-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of healthcare providers by evaluating how much diagnosis and management of neonatal shock adherent to Assuit University Children Hospital guidelines. | Baseline
  analysis of results and compare them to guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Safwat M Abd Al-ziz, lecture, Principal Investigator — Safwatabdelaziz371@yahoo.com

REFERENCES:
- [Background] Bhat BV, Plakkal N. Management of Shock in Neonates. Indian J Pediatr. 2015 Oct;82(10):923-9. doi: 10.1007/s12098-015-1758-7. Epub 2015 May 21. PMID 25990594
- [Background] de Boode WP, van der Lee R, Horsberg Eriksen B, Nestaas E, Dempsey E, Singh Y, Austin T, El-Khuffash A; European Special Interest Group 'Neonatologist Performed Echocardiography' (NPE). The role of Neonatologist Performed Echocardiography in the assessment and management of neonatal shock. Pediatr Res. 2018 Jul;84(Suppl 1):57-67. doi: 10.1038/s41390-018-0081-1. PMID 30072807
- [Background] Osborn DA, Evans N. Early volume expansion versus inotrope for prevention of morbidity and mortality in very preterm infants. Cochrane Database Syst Rev. 2001;2001(2):CD002056. doi: 10.1002/14651858.CD002056. PMID 11406028
- [Background] Ng PC, Lee CH, Bnur FL, Chan IH, Lee AW, Wong E, Chan HB, Lam CW, Lee BS, Fok TF. A double-blind, randomized, controlled study of a "stress dose" of hydrocortisone for rescue treatment of refractory hypotension in preterm infants. Pediatrics. 2006 Feb;117(2):367-75. doi: 10.1542/peds.2005-0869. PMID 16452355
- [Background] Femitha P, Bhat BV. Early neonatal outcome in late preterms. Indian J Pediatr. 2012 Aug;79(8):1019-24. doi: 10.1007/s12098-011-0620-9. Epub 2011 Dec 10. PMID 22161578
- [Background] Saugstad OD, Aune D. Optimal oxygenation of extremely low birth weight infants: a meta-analysis and systematic review of the oxygen saturation target studies. Neonatology. 2014;105(1):55-63. doi: 10.1159/000356561. Epub 2013 Nov 15. PMID 24247112
- [Background] Brierley J, Carcillo JA, Choong K, Cornell T, Decaen A, Deymann A, Doctor A, Davis A, Duff J, Dugas MA, Duncan A, Evans B, Feldman J, Felmet K, Fisher G, Frankel L, Jeffries H, Greenwald B, Gutierrez J, Hall M, Han YY, Hanson J, Hazelzet J, Hernan L, Kiff J, Kissoon N, Kon A, Irazuzta J, Lin J, Lorts A, Mariscalco M, Mehta R, Nadel S, Nguyen T, Nicholson C, Peters M, Okhuysen-Cawley R, Poulton T, Relves M, Rodriguez A, Rozenfeld R, Schnitzler E, Shanley T, Kache S, Skippen P, Torres A, von Dessauer B, Weingarten J, Yeh T, Zaritsky A, Stojadinovic B, Zimmerman J, Zuckerberg A. Clinical practice parameters for hemodynamic support of pediatric and neonatal septic shock: 2007 update from the American College of Critical Care Medicine. Crit Care Med. 2009 Feb;37(2):666-88. doi: 10.1097/CCM.0b013e31819323c6. PMID 19325359
- [Background] Osborn DA, Evans N. Early volume expansion for prevention of morbidity and mortality in very preterm infants. Cochrane Database Syst Rev. 2004;2004(2):CD002055. doi: 10.1002/14651858.CD002055.pub2. PMID 15106166
- [Background] Subhedar NV, Shaw NJ. Dopamine versus dobutamine for hypotensive preterm infants. Cochrane Database Syst Rev. 2003;(3):CD001242. doi: 10.1002/14651858.CD001242. PMID 12917901
- See also: pupmed — http://www.ncbi.nlm.nih.gov/pubmed/25990594
- See also: pupmed — http://www.ncbi.nlm.nih.gov/pubmed/11406028?dopt=Abstract